CLINICAL TRIAL: NCT04446793
Title: An Expanded Access Program of Onvansertib in Combination With FOLFIRI and Bevacizumab for the Second-Line Treatment of Patients With KRAS-Mutated Metastatic Colorectal Cancer (mCRC)
Brief Title: Expanded Access of Onvansertib With FOLFIRI and Bevacizumab for the Second-Line Treatment of Participants With KRAS-Mutated Metastatic Colorectal Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Other Study IDs: CRDF-01E
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Colorectal Cancer; KRAS Gene Mutation
Keywords: Colorectal Cancer; KRAS-Mutation; Onvansertib; PCM-075; FOLFIRI; Irinotecan; 5-Fluoruracil; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — onvansertib; Bevacizumab; IFL protocol

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Onvansertib — 15 mg/m^2 will be administered orally on Day 1 to Day 5 of every 14 day treatment course. There will be two 14-day courses of treatment in each 28 day cycle.
Biological: Bevacizumab — 5 mg/kg will be administered intravenously on Day 1 of every 14 day treatment course. There will be two 14-day courses of treatment in each 28 day cycle.
Drug: FOLFIRI — FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil [5-FU], and 2400 mg/m^2 continuous intravenous infusion 5-FU over 46 hours) will be administered intravenously on Day 1 of every 14 day treatment course. There will be two 14-day courses of treatment in each 28 day cycle.

SUMMARY:
This is an expanded access program for eligible participants designed to provide access to onvansertib in combination with FOLFIRI and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Participant is NOT eligible for other clinical trials currently open in the region
* Participant has failed or progressed on standard of care systemic therapy
* FOLFIRI (with or without 5FU bolus and continuous infusion)/bevacizumab plus onvansertib is appropriate for the participant as determined by the treating physician, including participants who have previously been treated with FOLFIRI
* Histologically confirmed metastatic and unresectable CRC with a confirmed KRAS mutation
* Age ≥ 18 years
* Participant was previously enrolled in an existing Cardiff clinical trial that is ending and based on investigator judgement has responded to treatment using onvansertib plus FOLFIRI (with or without 5FU bolus) + bevacizumab

Women of Child-bearing Potential

* Women of child-bearing potential (WOCBP) must agree to use method(s) of contraception
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of onvansertib treatment
* If sexually active, the participant must agree to use contraception considered adequate and appropriate by the treating physician during the period of onvansertib administration

Exclusion Criteria:

* Participant has not recovered from minor or major surgery and less than 6 weeks out from major surgery
* Participant has active Hepatitis B or C infection
* Participant has a known history of testing positive for human immunodeficiency virus or having been diagnosed with acquired immunodeficiency syndrome
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure Class II or higher according to the New York Heart Association Functional Classification, unstable angina pectoris, significant pulmonary disease (shortness of breath at rest or mild exertion), that would limit compliance with study requirements
* Abnormal glucuronidation of bilirubin, known Gilbert's syndrome
* Participants with any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the treating physician, would substantially increase risk to their well-being
* Any condition that, in the opinion of the treating physician, would substantially increase risk to their well-being

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult